CLINICAL TRIAL: NCT00231062
Title: Clinical Evaluation to Confirm Safety and Efficacy of Sinuplasty in the Paranasal Sinuses (CLEAR)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Integra LifeSciences Corporation (Industry)
Collaborators: Acclarent (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-00313
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Results first posted 2011-07-08 (Estimated); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Chronic Sinusitis
Keywords: sinusitis; rhinitis; sinus surgery; maxillary; ethmoid; sphenoid; frontal; FESS; sinuplasty
MeSH Terms: conditions — Sinusitis; Rhinitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Sinuplasty

SUMMARY:
A multi-center, non-randomized, prospective post-market evaluation of sinuplasty in paranasal sinuses.

DETAILED DESCRIPTION:
Sinusitis is a common healthcare problem that significantly reduces quality of life for people around the world. Patients suffer from headache, facial discomfort, nasal congestion, nasal drainage, loss of the sense of smell and malaise. Sinusitis is responsible for major healthcare expenditure and loss of workplace productivity.

The rationale of this study is to collect data on the effectiveness and safety of balloon dilation of the Frontal, Maxillary and Sphenoid sinuses by treating patients and observing them for a six month period of time following the procedure. Six month follow-up data is important to demonstrate the effectiveness of balloon catheter dilation.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and greater
2. Both male and female patients eligible
3. Diagnosis of chronic sinusitis that is not responsive to medical management
4. Planned endoscopic sinus surgery (recommended by PI, consented to by patient)

Exclusion Criteria:

1. Extensive sinonasal polyps
2. Extensive previous sinonasal surgery
3. Extensive sinonasal osteoneogenesis
4. Cystic fibrosis
5. Sampter's Triad (Aspirin sensitivity, Asthma, Sinonasal polyposis)
6. Sinonasal tumors or obstructive lesions
7. History of facial trauma that distorts sinus anatomy and precludes access to the sinus ostium
8. Ciliary dysfunction
9. Pregnant females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2005-04; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Church, MD, Principal Investigator — Loma Linda University

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from 3/2005 to 12/2005 in physician practice
Period: Overall Study
Arm/Group | Balloon Dilation of Sinus Ostia
Started | 115
Completed | 109
Not Completed | 6
Not completed — Physician Decision | 6

BASELINE CHARACTERISTICS:
Arm/Group | Balloon Dilation of Sinus Ostia
Number analyzed (Participants) | 115
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 102
  >=65 years | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (12.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74
  Male | 41
Region of Enrollment [Number; unit: participants]
  United States | 115

OUTCOME MEASURES:

1. Primary Outcome: Number of Sinuses With Patency of Sinus Ostium After Sinuplasty
Description: Patency of sinus ostium after sinuplasty will be determined by nasal endoscopic examination. The investigator will make a clinical judgment as to whether or not this has been achieved.
Time Frame: 24 weeks
Population: Analysis per Protocol; based on all sinuses of subjects not lost to follow-up at 24 weeks
Measure: Number; unit: Sinuses
Units Other Than Participants: sinuses
Arm/Group | Balloon Dilation of Sinus Ostia
Number analyzed (Participants) | 95
Number analyzed (sinuses) | 304
Sinuses | 247

2. Primary Outcome: Number of Participants With Adverse Events Following Sinuplasty Procedure
Description: Adverse event rate at 24 weeks: comprised of all observed peri-operative adverse events which were recorded on dedicated CRFs and any observed or patient-reported post-operative adverse events will be similarly recorded (through 24 week follow-up).
Time Frame: 24 weeks
Population: Analysis per protocol; based on subjects not lost to follow-up at 24 weeks
Measure: Number; unit: Participants
Arm/Group | Balloon Dilation of Sinus Ostia
Number analyzed (Participants) | 109
Participants | 9

3. Secondary Outcome: Number of Participants Experiencing Relief of Sinus Symptoms
Description: To gain general insight into the ability of balloon catheter sinus ostial dilation to relieve sinus symptoms, scores from the pre-operative SNOT-20 evaluations were compared to scores from the post-procedure SNOT-20 evaluations at 24 weeks following the procedure. The number of participants who showed aggregate symptom relief are recorded here as having been successfully treated.
Time Frame: Week 24
Population: All patients treated per protocol; includes all subjects not lost to follow-up at 24 weeks and who completed symptom questionnaire
Measure: Number; unit: Participants
Arm/Group | Balloon Dilation of Sinus Ostia
Number analyzed (Participants) | 95
Participants | 80

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Balloon Dilation of Sinus Ostia
Serious Adverse Events (participants affected / at risk) | 0/109
Other Adverse Events (participants affected / at risk) | 9/109
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Balloon Dilation of Sinus Ostia (N=109)
bacterial sinusitis (General disorders) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If requested by Sponsor, Investigator(s) shall delay the submission of any publication or presentation for up to sixty (60) days from the date of Sponsor's request to permit the preparation and filing of related patent applications by Sponsor or for Sponsor to take other steps to protect its intellectual property interests.